CLINICAL TRIAL: NCT05098600
Title: The Epidemiology, Management and Associated Conditions in Alopecia Areata in Czech Republic: A University-clinic-based Cross-sectional and Cohort Study
Brief Title: The Epidemiology, Management and Comorbidities in Alopecia Areata in Czech Republic
Status: Completed | Type: Observational
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Athanasios J. Stefanis, Prinicipal Investigator, Faculty Hospital Kralovske Vinohrady
Other Study IDs: NKS1001
Record Dates: First submitted 2021-10-16; First posted 2021-10-28 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis; Alopecia Areata (& Ophiasis); Alopecia Barbae; Alopecia Diffuse; Autoimmune Diseases; Autoimmune Hyperthyroidism; Autoimmune Hypothyroidism; Diabetes Mellitus, Type 1; Ulcerative Colitis; Inflammatory Bowel Diseases; Crohn Disease; Rheumatoid Arthritis; Down Syndrome; Atopic Dermatitis; Atopic Asthma; Atopic Rhinitis; Vitiligo; Psoriasis; Ankylosing Spondylitis; Multiple Sclerosis; Lupus Erythematosus; COVID-19 Pandemic; Vaccine Reaction; Infections; Anemia, Pernicious
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis; Diffuse alopecia; Autoimmune Diseases; Graves Disease; Hypothyroidism, Autoimmune; Diabetes Mellitus, Type 1; Colitis, Ulcerative; Inflammatory Bowel Diseases; Crohn Disease; Arthritis, Rheumatoid; Down Syndrome; Dermatitis, Atopic; Rhinitis, Allergic, Perennial; Vitiligo; Psoriasis; Spondylitis, Ankylosing; Multiple Sclerosis; COVID-19; Infections; Anemia, Pernicious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients with a confirmed histologic/dermatoscopic diagnosis of Alopecia areata within the study period will be included for analysis.
  Interventions: Other: Exposure of interest

INTERVENTIONS:
Other: Exposure of interest — Common autoimmune and atopic conditions consist of atopic dermatitis, allergic rhinitis, asthma, Crohn's disease, ulcerative colitis, Celiac disease, Pernicious anaemia, Type 1 diabetes, Autoimmune thyroiditis (Hashimoto's thyroiditis, Grave's disease, atrophic, unspecified), rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, polymyalgia rheumatica, Systemic lupus erythematosus, Sjogren syndrome, psoriasis, vitiligo, Multiple sclerosis

SUMMARY:
The study series consists of three studies with the aim to assess the incidence, prevalence, risk factors, comorbidities and management of patients with alopecia areata in Czech Republic based on the patients and registry of a dermatology clinic of a metropolitan hospital.

DETAILED DESCRIPTION:
The first study will aim to identify the incidence and prevalence of alopecia areata in the dermatology clinic of a metropolitan teaching hospital between 1/1/2011 and 31/12/2020

The second study will assess (1) the epidemiology of autoimmune and atopic diseases in patients with alopecia areata, (2) the presence of possible risk factors responsible for the onset/relapse/exacerbation of alopecia areata, (3) the levels of vitamin D and various autoantibodies,particularly thyroid autoantibodies and (4) the variety, duration, efficacy and safety profile of treatment modalities used in our hospital for the management of alopecia areata from 15/10/2021 to 14/10/2022.

The third study will monitor the monthly oscillations of vitamin D and thyroid-autoantibodies of patients with new-onset/relasping or exacerbating alopecia areata for six months, between 15/10/2021-14/10/2022 in order to observe if changes in levels of vitamin D and thyroid-antiantibodies are associated with severity and prognosis (worsening or improvement) of alopecia areata

ELIGIBILITY:
Inclusion Criteria:

* All patients visiting our clinic with a dermatologic condition between 1/1/2011-31/12/2020
* For the second study, only patients with histologic/dermatoscopic diagnosis of new-onset/relapsing/peristent-untreated alopecia areata, presenting to our clinic between 15/10/2021-14/10/2022 are included.

Exclusion Criteria:

* For the second study patients with other alopecias, patients denying data sharing despite signing the informed concent and presenting outside the study period are excluded.
* For the third study, patients with other types of alopecia, as well as those who signed the informed consent but refused to share their data or undergo blood tests at our hospital, and those who did not visit our outpatient department at least once a month for the required duration, were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and children patients with a dermatologic condition between 1/1/2011-31/12/2020 and for the second study, adults and children with first-onset/relapsing/persistent-untreated alopecia areata visiting our clinic between 15/10/2021 and 14/10/2022 who sign informed consent are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
The epidemiology of Alopecia areata | 1/1/2011-31/12/2020
  The incidence and point prevalence of Alopecia areata within the study cohort during the study period, stratified by age-group and gender
The epidemiology of Alopecia areata | 1/10/2020-30/9/2021
  The incidence and point prevalence of Alopecia areata (totalis, universalis, ophiasis, sisaipho, reticularis, diffuse, barbae) within the study cohort during the study period, stratified by age-group and gender
Prevalence of atopic and autoimmune conditions in patients with Alopecia Areata | 15/10/2021-14/10/2022
  Prevalence of atopic and autoimmune conditions in patients with Alopecia Areata
Treatments for alopecia areata | 15/10/2021-14/10/2022
  Assessment of various treatment modalities used for alopecia areata
Safety and efficacy of treatments in alopecia areata | 15/10/2021-14/10/2022
  Assessment of various treatment modalities used for alopecia areata, efficacy, duration of treatment, reported side-effects and relapse rate after withdrawal
Measurement of Thyroid stimulating hormone (TSH) | 15/10/2021-14/10/2022
  Measurement of TSH on first visit and once a month for 6 months. Normal values for adults 0.550-4.780 mu/l according to our laboratory. All blood tests will be performed in our laboratory at the day of the visit before any clinical examination
Measurement of free Thyroxine (fT4) | 15/10/2021-14/10/2022
  Measurement of fT4 on first visit and once a month for 6 months. Normal values for adults 11.50-22.70 pmol/l according to our laboratory. All blood tests will be performed in our laboratory at the day of the visit before any clinical examination
Measurement of free Triodothyronine (fT3) | 15/10/2021-14/10/2022
  Measurement of fT3 on first visit and once a month for 6 months. Normal values for adults 3.50-6.50 pmol/l according to our laboratory. All blood tests will be performed in our laboratory at the day of the visit before any clinical examination
Measurement of Thyroid peroxidase autoantibodies (TPOAbs) | 15/10/2021-14/10/2022
  Measurement of TPOAbs on first visit and once a month for 6 months. Normal values for adults <60 kU/l according to our laboratorypmol/l. All blood tests will be performed in our laboratory at the day of the visit before any clinical examination
Measurement of thyreoglobulin autoantibodies (TgAbs) | 15/10/2021-14/10/2022
  Measurement of TgAbs on first visit and once a month for 6 months. Normal values for adults <4.5 kIUl/l according to our laboratory. All blood tests will be performed in our laboratory at the day of the visit before any clinical examination
Measurement of anti TSH receptor antibodies (TRAbs) | 15/10/2021-14/10/2022
  Measurement of TRAbs on first visit and once a month for 6 months. Normal values for adults <1.22 Ul/l according to our laboratory. All blood tests will be performed in our laboratory at the day of the visit before any clinical examination
Measurement of Vitamin D levels | 15/10/2021-14/10/2022
  Measurement of Vitamin D levels on first visit and once a month for 6 months. Normal values for adults are 75.0-250.0 nmol/l acording to our laboratory. All blood tests will be performed in our laboratory at the day of the visit before any clinical examination

SECONDARY OUTCOMES:
Prevalence of atopic and autoimmune conditions in the family history of patients with Alopecia Areata | 15/10/2021-14/10/2022
  Prevalence of atopic and autoimmune conditions in parents and siblings of patients with Alopecia Areata
Identification and prevalence of possible exacerbating factors in patients with Alopecia Areata | 15/10/2021-14/10/2022
  Identification of possible risk factors occuring within 6 months from the onset/relapse/worsening of alopecia areata, according to patient history

CONTACTS AND LOCATIONS:
Locations (1):
- Teaching Hospital of Royal Vineguards, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided